CLINICAL TRIAL: NCT03207464
Title: Molecular Imaging of Norepinephrine Transporter (NET) Using [C-11]Methylreboxetine PET in Multiple Sclerosis
Brief Title: Molecular Imaging of NET Using [C-11]MRB-PET in MS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, TARUN SINGHAL, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P001099
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple Sclerosis (Experimental): Subjects meeting the definition for Multiple Sclerosis by the International Panel Criteria, with an Expanded Disability Status Scale (EDSS) less than 6.5.
  Interventions: Drug: [C-11]Methylreboxetine
- Healthy Control (Experimental): This group will serve as non disease population.
  Interventions: Drug: [C-11]Methylreboxetine

INTERVENTIONS:
Drug: [C-11]Methylreboxetine — 8 individuals with Multiple Sclerosis and 4 healthy controls will undergo a [C-11]MRB PET scan and a MRI scan.
  Other Names: [C-11]MRB

SUMMARY:
This study aims to use [C-11]MRB PET (positron emission tomography) imaging to look at brain injury in patients with Multiple Sclerosis (MS) and healthy individuals. The overarching hypothesis is that there is decreased radioligand binding to the norepinephrine transporter in multiple sclerosis, reflecting injury to the noradrenergic system and that it plays a role in disease pathogenesis, its clinical manifestations and severity. This strategy is targeted to address an unmet need because currently available MRI techniques lack sensitivity and specificity for assessing such changes in the brains of people with MS.

The specific aims of the study are:

1. To determine norepinephrine transporter binding in the brains of MS patients using [C-11]MRB PET and compare it with age, and sex matched healthy controls.
2. To determine correlation of norepinephrine transporter binding with clinical severity and MRI parameters in MS.
3. To determine correlation of norepinephrine transporter binding with fatigue and cognitive impairment in MS patients.

DETAILED DESCRIPTION:
Two groups of subjects will be recruited:

1. Individuals meeting the definition for Multiple Sclerosis by the International Panel Criteria19, with an Expanded Disability Status Scale (EDSS) less than 6.5
2. Age- and sex-matched healthy controls

The goal sample size is 12 subjects including 4 healthy controls and 8 subjects with Multiple Sclerosis (MS).

Subjects will be recruited by the PI, one of the other co-investigators, or a staff member listed on the protocol at the Partners MS Center and the Behavioral Neurology Clinic of Brigham and Women's Hospital.

Side Effects Monitoring:

No side effects from the radiopharmaceutical are expected nor have they been reported with C-11 MRB. As this study is conducted under MGH (Massachusetts General Hospital) RDRC (Radioactive Drug Research Committee) oversight, the administered dose of C-11 MRB is well below the known level to cause any pharmacologic effect. Subjects will also be exposed to a small amount of radiation.

Subject Safety:

Subject monitoring during MRI and PET scans will be performed using a 2-way intercom system between the scanner operator and subject and by visual monitoring of the subject through the window into the scan room (the subject is visible to the operator at all times).

Subjects will need to lie still in the PET camera for period of 120 min, and subjects may find it uncomfortable to remain still over this time. Therefore, as mentioned above, subjects will be given the opportunity to take a break for up to 20 minutes after 70 minutes of PET scanning, following which the last 30 minutes of scanning will be completed. A standard head-support device will be used to make the subjects comfortable during the scanning.

If subjects find an arterial line or duration of scanning too uncomfortable, they are free to withdraw from the study at any time.

The MRI scans take place in a confined space that makes some people claustrophobic. Claustrophobic individuals will be excluded from the study. Also during the scan the subject will hear loud banging noises and will therefore wear ear plugs to reduce this noise.

Recruitment Process:

Physicians at the Partners MS Center and the Brigham and Women's Hospital (BWH) Behavioral Neurology clinic may present the study to a subject during a regular scheduled clinic visit. If the subject is interested in the study, a copy of the consent form will be given. At the time of the subject's initial screening visit, a licensed physician investigator will answer any questions the subject may have regarding the study and subsequently obtain informed consent. In accordance with NIH guidelines, efforts will be made to attain a mix of study participants, in terms of gender and racial/ethnic representation.

Consent Process:

Informed consent will be obtained from the subjects by a licensed physician investigator on the study protocol. If the investigator is a clinician from the MS Center clinic, they will not be allowed to obtain consent from their own patients. Existing MS Center subjects may be sent a letter describing the study and a copy of the consent document. Interested subjects are directed to contact research staff via a telephone number provided in the letter inviting participation in the study to set up a screening visit. They will have the opportunity to discuss the study with research study staff prior to giving consent as outlined above. Subjects approached for participation in the study during a routine clinical visit will have the opportunity to participate in the study at that time or they may choose to return for participation at another time in the future. All subjects will be informed that they are free to withdraw consent from the study at any time without affecting the quality or type of care that they receive at BWH or MGH.

Monitoring and Quality Assurance:

During the study period, subjects will be followed by their clinical neurologists for adverse events and disease progression. If problems are reported to their physicians, they will receive care as is normally performed. In addition, the Principal Investigator (PI) will review all laboratory results of tests undergone by the subjects during the study period and help co-ordinate any necessary care with patient's primary providers.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals meeting the definition for Multiple Sclerosis by the International Panel Criteria, with an Expanded Disability Status Scale (EDSS) less than 7.5
2. Male and female subjects age 18 to 70 years
3. Subjects willing to undergo PET and MRI imaging
4. Subjects willing and able to give informed consent

Exclusion Criteria:

1. Individuals with a comorbid severe psychiatric condition such as schizophrenia, bipolar disorder, or post-traumatic stress disorder.
2. Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
3. Individuals taking tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors, or norepinephrine-dopamine reuptake inhibitors.
4. Concurrent medical conditions that contraindicate study procedures.
5. Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
6. Claustrophobia
7. Non-MRI compatible implanted devices
8. Corticosteroid treatment in the past four weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
[C-11]Methylreboxetine area under the curve ratios | Baseline
  PET Imaging measurement

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham MS Center, 60 Fenwood Road, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No